CLINICAL TRIAL: NCT02417259
Title: Changes in Cerebral and Somatic Near Infrared Spectroscopy Monitoring Before and After Surgery for in Children With Cyanotic Heart Disease
Brief Title: Near Infrared Spectroscopy in Cyanotic Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Covidien Private Limited (Unknown)
Responsible Party: Principal Investigator, Judith Wong Ju-Ming, MBBCh BAO, MRCPCH, KK Women's and Children's Hospital
Other Study IDs: 2015/2161
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Congenital Heart Defects
Keywords: Spectroscopy, Near-Infrared
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We are conducting a prospective cohort study of 20 children with cyanotic congenital heart disease who are admitted for cardiac surgery. We will record cerebral and somatic near infrared spectroscopy (NIRS) at two sites - forehead and flank regions using the Covidien INVOS™ 5100C Cerebral / Somatic Oximeter. The monitoring will begin one hour pre-operatively (baseline) and continue until 48hours post-operatively. We will also take measurements prior to discharge from hospital. Baseline demographics, physiological and laboratory variables will be recorded. Clinical outcome variables including mortality, duration of intensive care unit (ICU) stay, duration of mechanical ventilation, inotropic support and feed tolerance will also be recorded.

DETAILED DESCRIPTION:
NIRS has been used to predict short term clinical outcomes (low cardiac output states, prolonged ventilation, and prolonged hospital stay) and long term clinical outcomes (reduced neurodevelopmental scores at 1year, radiological changes on magnetic resonance imaging). NIRS has also been tested against traditional markers of global tissue perfusion like mixed venous saturation and serum lactate, however, results from these studies are mixed. There is insufficient prospective data evaluating NIRs with direct clinical outcomes and uncertainty about the threshold value or the duration below a threshold value that leads to tissue injury. Because of this lack of data, the benefit and risk of management strategies targeted to improve NIRS values remains unknown.

We will characterize the time series of cerebral and somatic oximetry, pulse oximetry and partial pressure of arterial oxygen in the cyanotic child undergoing surgical repair of a congenital heart defect. We will then determine the correlation between the time series if any. This new information will advance our understanding of the hemodynamic changes that occur in the perioperative period and may lead to new therapeutic targets.

The primary hypothesis is that there is a delayed increase in cerebral and somatic oximetry post-operation as compared pulse oximetry (SpO2) and partial pressure of arterial oxygen (PaO2) which occur immediately.

The secondary hypothesis is to establish the applicability of a desaturation score (decrease of 20% in area under the curve [AUC] over an hour) in the early prediction of adverse outcomes.

The oximetry probes will be placed pre-induction of anesthesia (to determine baseline) and recordings will be continuous throughout the operation and 48hours post-operatively. Children undergoing cardiac surgery generally stay in the hospital for 1-2weeks. We will also take oximetry measurements prior to discharge from hospital (to determine the new steady state). Sites measured are cerebral (forehead) and somatic (left flank).

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative diagnosis of cyanotic congenital heart disease
* Undergoing any form of cardiac surgery
* Informed consent was given by the caregiver/parent

Exclusion Criteria:

* Premature infants <35 weeks corrected age who will be cared for in the neonatal ICU postoperatively
* Congenital lactic acidosis syndromes

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cyanotic congenital heart disease undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in cerebral oximetry | 48horus post-operatively
  To show if there is a delayed increase in cerebral oximetry post-operation as compared SpO2 and PaO2 which occur immediately
Change in somatic oximetry | 48hours post-operatively
  To show if there is a delayed increase in somatic oximetry post-operation as compared SpO2 and PaO2 which occur immediately

SECONDARY OUTCOMES:
Applicability of a desaturation score in the early detection of adverse outcomes | 48hours post-operatively
  Cerebral desaturation score (>20% decrease in AUC over an hour) for early detection of adverse outcome such as cardiorespiratory deterioration requiring chest tube insertion, re-do surgery, chest compressions, electrical shock or initiation of extracorporeal membrane oxygenation.

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Bukit Timah Road, Singapore, Singapore

REFERENCES:
- [Derived] Wong JJ, Chen CK, Moorakonda RB, Wijeweera O, Tan TYS, Nakao M, Allen JC Jr, Loh TF, Lee JH. Changes in Near-Infrared Spectroscopy After Congenital Cyanotic Heart Surgery. Front Pediatr. 2018 Apr 13;6:97. doi: 10.3389/fped.2018.00097. eCollection 2018. PMID 29707528